CLINICAL TRIAL: NCT04976335
Title: Quantitative and Clinical Assessment of Flexor Tendon Gliding Following Application of a Bioresorbable Hydrogel: A Prospective, Randomized Study in Patients Undergoing Distal Radius Fracture Repair.
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Prevention
Other Study IDs: 20-2659
Record Dates: First submitted 2021-07-14; First posted 2021-07-26 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Distal Radius Fracture; Tendon Rupture
MeSH Terms: conditions — Wrist Fractures

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (2):
- Versawrap (Active Comparator)
  Interventions: Device: Versawrap membrane
- No Versawrap (No Intervention)

INTERVENTIONS:
Device: Versawrap membrane — Versawrap membrane will be placed between distal radius plate and flexor tendons
  Arms: Versawrap

SUMMARY:
The investigators will be evaluating the use of versawrap in the setting of distal radius fractures by placing membrane between plate and flexor tendons. Investigators will then evaluate tendon gliding morphology and number of tendon ruptures

ELIGIBILITY:
Inclusion Criteria:

* Cognitively able to converse in English or in native language supported by a certified medical interpreter;
* Diagnosed with a closed, distal radius fracture treated with open reduction and internal fixation using a volar distal radius plating system.

Exclusion Criteria:

* open injury;
* concomitant injury to the contralateral wrist;
* history of flexor tendon repair involving one or both hands or wrists;
* use of a trans-carpal fixation device (bridge plate or external fixator) that would preclude wrist motion post-operatively;
* concomitant fracture / injury to the thumb or index finger of one or both hands;
* concomitant carpal tunnel release.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-09-13 (Actual); Primary Completion 2027-07 (Estimated); Study Completion 2027-07 (Estimated)

PRIMARY OUTCOMES:
Range of Motion: Thumb Interphalangeal and Index Finger Distal Interphalangeal Joints | 6 months
  Standardized clinical examination (relative to wrist and digital positioning): active and passive range of motion for thumb interphalangeal and index finger distal interphalangeal joints.
Range of Motion: Thumb and Index Finger | 6 months
  Standardized clinical examination (relative to wrist and digital positioning): active and passive composite digital range of motion for thumb and index fingers
Range of Motion: Wrist | 6 months
  Standardized clinical examination (relative to wrist and digital positioning): active and passive wrist range of motion.
Ultrasound Assessment of Flexor Pollicis Longus and Index Finger Flexor Digitorum Profundus Tendon Excursion | 6 Months
  Tendons in the volar forearm will be directly visualized with ultrasound. The distance the tendons are able to travel (excursion) within the forearm will be reported.

SECONDARY OUTCOMES:
Complications | 6 months
  Incidence of any of the following perioperative complications: infection, neurovascular injury, tendon rupture, hardware failure, delayed fracture union, fracture nonunion, fracture malunion, or revision surgery
Patient-Rated Wrist Evaluation (PRWE) | 6 Months
  The Patient-Rated Wrist Evaluation (PRWE) measures pain and wrist function. Possible scores range from 0-100, with a higher score indicating a worse outcome.
Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) | 6 Months
  The Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) measures limb function and disability. Possible scores range from 0-100, with a higher score indicating a worse outcome (more severe disability).
Visual Analog Scale (VAS) pain scores | 6 Months
  The Visual Analog Scale measures patient reported pain using a 100mm scale. Possible scores range from 0-100, with higher scores indicating more severe pain.
Subjective Reporting Specific to Tendon Function | 6 Months
  The number of participants reporting the following: 1) pain with resist pinch, 2) perceived tendon triggering, catching, or locking
Ultrasound Assessment of Flexor Pollicis Longus and Index Finger Flexor Digitorum Profundus Tendon Morphology | 6 Months
  Tendons in the volar forearm will be directly visualized with ultrasound and their physical appearance will be grossly described. For this outcome measure, the number of participants with a healthy tendon, as determined by the physician, will be reported.
Key Pinch | 6 Months
  Standardized clinical examination (relative to wrist and digital positioning) of key pinch.
Three-Jaw Pinch | 6 Months
  Standardized clinical examination (relative to wrist and digital positioning of three-jaw pinch.
Grip Strength | 6 Months
  Standardized clinical examination (relative to wrist and digital positioning) of grip strength.
Soong Classification | 6 Months
  Routine (3-view) radiographs of the injured wrist to document Soong grading of distal radius plate positioning. Soong et al (2011) proposed the Soong classification to classify palmar prominence at the watershed line, where flexor tendons lie closest to the plate. Classifications are as follows: 0: Plates do not extend volar to the watershed line; 1: Plates are volar to the line, but proximal to the volar rim; and 2: Plates are directly on or distal to the volar rim.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - University of Colorado Health Hospital, Aurora, Colorado
  - Denver Health Hospital, Denver, Colorado

IPD SHARING:
Plan to Share IPD: No